CLINICAL TRIAL: NCT05601037
Title: Lymfo-Veneuse Anastomosen Ter Preventie Van Lymphoedeem
Brief Title: LymphoVenous Anastomosis to Prevent Breast Cancer Related Lymphedema
Acronym: LVARCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BC-09374; 2021-004751-16 (EudraCT Number)
Record Dates: First submitted 2021-11-09; First posted 2022-11-01 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Lymphedema, Breast Cancer
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: blinded randomized prospective
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Axilla dissection + Lymphevenous Anastomosis (Experimental): Surgical bypass between lymphatic vessel and vein
  Interventions: Procedure: Axilla dissection + Lymphovenous anastomosis
- Standard surgery (No Intervention): Standard surgery

INTERVENTIONS:
Procedure: Axilla dissection + Lymphovenous anastomosis — surgical bypass between lymphatic vessel and vein
  Arms: Axilla dissection + Lymphevenous Anastomosis

SUMMARY:
Lymphedema is defined as a chronic condition, caused by lymphostasis. A major part in the Western world consists of iatrogenic lymphedema caused by surgery to the lymph nodes of the axilla or groin. Prophylactic lymphovenous anastomosis (LVA) could be beneficial in the prevention of lymphedema of the extremities.

DETAILED DESCRIPTION:
The investigator is performing a blinded randomized prospective study on 80 patients undergoing an axilla dissection for their breast cancer treatment. One group will receive a LVA at the time of their axilla dissection. Other group will receive standard of care. Follow-up is 2 year.

ELIGIBILITY:
Inclusion Criteria:

* lymph node + breast cancer requiring dissection

Exclusion Criteria:

* previous lymphedema
* BMI >35

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
The volume via circumferential measurements: swelling < 5% | 2 years
  Comparing the volume of the arm at each study visit via circumferential measurements: swelling < 5%

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Depypere, MD, Principal Investigator — UZ GENT
Locations (1):
- UZ GENT, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Depypere B, Vyncke T, Dhooghe N, Claes K, Blondeel P, Van Landuyt K. A Novel Technique for Preventive Lymphovenous Anastomosis: Anastomosing a Ligated Lymphatic Vessel. Plast Reconstr Surg Glob Open. 2021 Mar 22;9(3):e3509. doi: 10.1097/GOX.0000000000003509. eCollection 2021 Mar. PMID 33968557